CLINICAL TRIAL: NCT05552677
Title: Effects of Multicomponent Training on Inflammation Parameters in Correlation With Muscle Quality and Function in Elderly Obese Woman
Brief Title: Effects of Multicomponent Training on Inflammation Parameters and Muscle Quality in Elderly Obese Woman
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ellen Cristini de Freitas, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Exercise_Inflammation
Record Dates: First submitted 2022-09-15; First posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Aging Disorder; Obesity; Inflammation
Keywords: anabolic resistance; obesity; inflammation; physical exercise
MeSH Terms: conditions — Obesity; Inflammation; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (CG) (No Intervention): Patients will recieve no intervention for the period of 12 weeks
- Exercise Group (EG) (Experimental): Patients will undergo a 12 week multicomponent training program
  Interventions: Other: Multicomponent Training

INTERVENTIONS:
Other: Multicomponent Training — Participants will perform a multicomponent training that explores strength, aerobic and balance capacities with load progression every 15 days. The sessions will last 60 minutes each, being held three times a week with a day of rest in between. The intervention will last 12 weeks
  Arms: Exercise Group (EG)

SUMMARY:
Population aging worldwide has increased substantially in recent years. In order to prevent disabling diseases and improve the quality of life, it is necessary to understand the conditions related to the health of this specific population. One of the known alterations that occur in the body is the increased low-grade systemic inflammatory process, anabolic resistance, and muscle catabolism. These conditions can negatively interfere with muscle quality and functionality. However, the maintenance of the metabolic and physical functionality of muscle tissue can be preserved by performing physical exercises throughout life because of its anti-inflammatory mechanisms. In the present study, a multicomponent training program that combines aerobic, strength, balance, and flexibility capacities was used. The hypothesis is that performing this type of physical exercise will mitigate meta-inflammation and its negative effects, in addition to stimulating anabolic signals and reducing insulin resistance present in anabolic resistance, leading to improved quality and muscle functionality in elderly women with obesity.

DETAILED DESCRIPTION:
Population aging worldwide has increased substantially in recent years. Therefore, it is necessary to know and understand the conditions related to the health of this specific population in order to prevent disabling diseases and improve the quality of life. One of the major concerns associated with the senescence process is the various physiological changes that can occur in the body. Body composition changes, bone loss, muscle catabolism, an increased low-grade systemic inflammatory process, and anabolic resistance all contribute to the development and/or worsening of several aging-related diseases. In particular, chronic low-grade inflammation, also known as meta-inflammation, can negatively interfere with muscle quality and functionality by reducing the muscle's ability to use energy substrates, amino acids, and perform protein synthesis. However, the maintenance of the metabolic and physical functionality of muscle tissue can be preserved by performing physical exercise throughout life because physical exercise can stimulate anti-inflammatory mechanisms. In the present study, a multicomponent training program will be used, which consists of training that combines aerobic, strength, balance, and flexibility capacities, and is capable of reducing inflammatory parameters and increasing physical and muscular capacities, resulting in a better quality of life and being thus attractive to this specific population. In view of this approach, the hypothesis is that performing this type of physical exercise is capable of mitigating meta-inflammation and its negative effects, in addition to stimulating anabolic signals and reducing insulin resistance present in anabolic resistance, leading to improved quality and muscle functionality in elderly women with obesity.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 30 and 40kg/m²;

Exclusion Criteria:

* alcoholics
* smokers
* diseases that prevents the practice of physical activity
* medical impediment to the practice of physical exercise throughout the study
* infectious diseases
* coronary diseases
* chronic kidney diseases
* chronic use of corticosteroids
* chronic use of immunomodulators
* undergoing nutritional monitoring or weight loss treatment
* score ≤13 for cognitive screening on the Mini-Mental State Examination (MMSE)

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 38 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in inflamatory markers | 12 weeks
  Evaluate the inflamatory markers PCR, IL-1β, IL-6, IL-10, IL-15, TNF-α, NFκβ, NLRP3, myonectin, SIRT1, sTNFR1, IL-10, IL-13, adiponectin
Changes in muscle quality | 12 weeks
  Evaluate the quantity of intramuscular fat deposits trough ultrasound pre and post intervention

SECONDARY OUTCOMES:
Changes in muscle function | 12 weeks
  Evaluate the muscle function trough the load test pre and post intervention
Changes in metabolic parameters - fasting blood glucose | 12 weeks
  Changes in fasting blood glucose samples in pre and post intervention
Changes in metabolic parameters - insulin sensitivity | 12 weeks
  Changes in insulin sensitivity, estimated through HOMA-IR pre and post intervention
Changes in muscle remodeling peptides | 12 weeks
  Changes in PNPLA3 and PNP3 in blood samples in pre and post intervention
Body composition changes | 12 weeks
  Changes in fat-free mass and fat mass evaluated pre and post intervention by iDEXA
Changes of physical performance | 12 weeks
  Physical performance changes, evaluated through physical tests.
Changes in blood myostatin | 12 weeks
  Changes in blood myostatin levels pre and post intervention
Indirect calorimetry assessment | 12 weeks
  Changes in resting metabolic rate (RMR) evaluated pre and post intervention by indirect calorimetry
Changes in metabolic parameters - lipid profile | 12 weeks
  Changes in lipid profile (total cholesterol, HDL-c, LDL-c, triglycerides)samples in pre and post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ellen C de Freitas, PhD, Principal Investigator — University of São Paulo, School of Physical Education and Sports of Ribeirão Preto.
Locations (1):
- University of São Paulo, School of Physical Education and Sports of Ribeirão Preto, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Travieso SG, Ortiz GU, Abud GF, Villalba MM, Junqueira GP, Gomes MM, Marchini JS, Freitas EC. Effects of Multicomponent Training on Metabolic and Functional Health of Older Women With Obesity: A Randomized Clinical Trial. J Aging Phys Act. 2025 Aug 26:1-13. doi: 10.1123/japa.2024-0341. Online ahead of print. PMID 40858281